CLINICAL TRIAL: NCT07190638
Title: Comparison of Outcomes and Surgical Time Between Cortical and Medullary Suture vs. Medullary-Only Suture: Cortex Clinical Trial, From 2025 to 2027
Brief Title: Comparison of Outcomes and Surgical Time Between Cortical and Medullary Suture vs. Medullary-Only Suture: Cortex Clinical Trial
Acronym: CORTEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Institute of Robotic Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 87015525.0.1001.5128
Record Dates: First submitted 2025-07-25; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: RCC, Renal Cell Cancer
Keywords: Partial Nephrectomy; Robot-assisted; MEDULLARY SUTURE; MEDULLARY-ONLY SUTURE
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: The first group will undergo medullary-only suturing (single-layer) using 3-0 diameter synthetic absorbable monofilament poliglecaprone 25 suture (Caprofyl™), with early unclamping performed robotically. In the second group, both medullary and cortical suturing (two-layer) will be performed, using 3-0 Caprofyl™ for the medullary suture and, after early unclamping, 0-diameter braided synthetic absorbable polyglycolic suture (Vicryl™) for the cortical layer, also robotically assisted.
  If the surgeon deems it necessary to perform a second suture using Vicryl™ 0 in the first group after unclamping, it will be carried out, and the surgeon's reasoning will be documented. These patients will be analyzed separately in order to identify predictive factors for such a change.
  Hemostatic agents will be used in all groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The blinding protocol will include the patient, the physician responsible for patient selection, the physician overseeing postoperative care, the professional conducting follow-up consultations, the students involved in collecting clinical follow-up data, and the team responsible for statistical analysis. However, the surgical team and the operating surgeon will not be blinded, nor will the students responsible for collecting intraoperative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medullary-only suturing (single-layer) (Experimental): After partial nephrectomy, only the medullary layer is sutured using a running 3-0 synthetic absorbable monofilament suture (Caproyl™). The cortical layer is not sutured. Hemostatic agents, such as Bleed Stp Plus, Surgicel® Fibrillar, or Hemopatch®, may be applied to support hemostasis.
  Interventions: Procedure: Medullary-only suturing (single-layer); Device: Suture; Device: Hemostatic Agent
- Medullary and cortical suturing (two-layer) (Active Comparator): After partial nephrectomy, both the medullary and cortical layers are sutured. The medullary layer is closed with a running 3-0 Caproyl™ suture before unclamping. Then, the cortical layer is sutured with 0 Vicryl™ using a running technique. Hemostatic agents, such as Bleed Stp Plus, Surgicel® Fibrillar, or Hemopatch®, may be applied to assist in bleeding control.
  Interventions: Procedure: Medullary and cortical suturing (two-layer); Device: Suture; Device: Hemostatic Agent

INTERVENTIONS:
Procedure: Medullary-only suturing (single-layer) — Only the base layer (medulla) is sutured after tumor excision, Cortical suturing is omitted. Hemostatic agents are applied.
  Other Names: Single-layer renorrhaphy
  Arms: Medullary-only suturing (single-layer)
Device: Suture — Synthetic absorbable monofilament suture (Caproyl™ 3-0).
  Arms: Medullary-only suturing (single-layer)
Procedure: Medullary and cortical suturing (two-layer) — Both medullary and cortical layers are sutured after tumor excision, Performed with robotic assistance using absorbable sutures. Hemostatic agents are applied
  Other Names: double-layer renorrhaphy
  Arms: Medullary and cortical suturing (two-layer)
Device: Suture — Synthetic absorbable monofilament suture (Caproyl™ 3-0), absorbable braided suture (Vicryl™ 0)
  Arms: Medullary and cortical suturing (two-layer)
Device: Hemostatic Agent — Hemostatic agents (e.g., Bleed Stp Plus, Surgicel® Fibrillar, Hemopatch®).

SUMMARY:
Renal function preservation is a growing concern in the surgical management of kidney tumors, particularly with the rise in chronic kidney disease worldwide. Recent surgical innovations have focused on modifying renorrhaphy techniques to minimize renal damage. Emerging evidence suggests that omitting cortical suturing may reduce operative time, blood loss, and renal parenchymal loss without increasing major complications. This randomized controlled trial aims to compare outcomes between medullary-only and combined cortical-medullary suture techniques during robot-assisted partial nephrectomy, with the goal of identifying the approach that best balances functional preservation and surgical safety.

DETAILED DESCRIPTION:
To investigate the clinical impact of a potentially modifiable surgical variable, namely, the choice of suture technique during renal reconstruction, on patient outcomes following robot-assisted partial nephrectomy.

The preservation of renal function has become a central concern in the surgical management of renal tumors, especially given the long-term consequences of chronic kidney disease on patient morbidity and mortality. Partial nephrectomy is preferred for localized renal masses as it allows for oncologic control while maintaining renal function. Traditionally, renorrhaphy involves a two-layer closure including both medullary and cortical sutures. However, recent literature suggests that omitting the cortical suture may reduce renal parenchymal volume loss and warm ischemia time, while possibly introducing a higher rate of minor complications.

Despite growing interest in minimally invasive nephron-sparing techniques, robust prospective and randomized trials directly comparing single-layer (medullary-only) and double-layer (cortical and medullary) renorrhaphy remain scarce. The single-layer technique, first proposed to address concerns over unnecessary cortical compression and ischemic injury, is gaining attention for its simplicity and potential advantages in reducing blood loss and operative time.

This trial aims to evaluate whether avoiding cortical suturing during robot-assisted partial nephrectomy leads to improved postoperative renal function, reduced blood loss, and shorter surgical duration. Patients will be randomly assigned to undergo either medullary-only renorrhaphy or the conventional dual-layer approach. Both techniques will be assessed for their effect on warm ischemia time, complication rates, renal volume loss, and surgical efficiency.

The study will enroll 80 patients undergoing partial nephrectomy for renal masses, distributed evenly across the two intervention groups. This sample size was calculated to ensure statistical power to detect differences in estimated blood loss, the primary outcome. A broad range of secondary outcomes will be measured at multiple postoperative time points, including estimated glomerular filtration rate, renal volume, incidence of surgical complications, and quality of life indicators.

By employing a randomized, prospective, and blinded design, the trial seeks to minimize bias and deliver high-quality evidence to guide future surgical decision-making. Ultimately, the study aims to clarify whether cortical renorrhaphy can be safely omitted without compromising patient outcomes, potentially simplifying surgical technique and improving recovery profiles in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of renal mass confirmed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Indication for partial nephrectomy
* Written informed consent
* Expected survival of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) score performance status ≤ 1
* Negative serum or urine pregnancy test within 24 hours before surgery for women of childbearing potential
* Recovery from any prior therapy-related toxicity to grade 1 or better
* If a biopsy has been performed, pathology consistent with renal cell carcinoma (RCC)

Exclusion Criteria:

* Solitary kidney
* Multiple or bilateral renal masses if more than one mass is operated on simultaneously or within less than 4 months
* Hepatic or renal toxicity grade ≥ 2 with glomerular filtration rate (GFR) < 30 according to Common Terminology Criteria for Adverse Events (CTCAE v4)
* Bleeding diathesis
* Inability to maintain anticoagulation for surgery
* Participation in another experimental trial simultaneously or within 30 days prior to enrollment
* Significant acute or chronic medical, neurological, or psychiatric condition that could compromise safety, limit study completion, or impair study objectives in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Estimated Blood loss | Perioperative/Periprocedural time
  Estimated blood loss, assessed to compare renorrhaphy techniques (single medullary suture vs. combined medullary and cortical suture) during partial nephrectomy. The volume, recorded in milliliters, was measured using a graduated collection canister connected to the assistant surgeon's suction device, with correction for the amount of saline solution instilled into the cavity.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) | 1 day, 2 weeks, 2 months, and 5 months
  Difference in eGFR values calculated using the CKD-EPI formula between baseline (preoperative) and postoperative time points
Percentage renal volume loss | 4 months
  Percentage reduction in renal parenchymal volume calculated from CT scan measurements at 4 months compared with baseline preoperative volume.
Warm ischemia time | Perioperative/Periprocedural time
  Duration, in minutes, of arterial clamping recorded during partial nephrectomy
Participants with intraoperative or postoperative complications | Through 5 months
  Number of participants experiencing complications such as hematuria, pseudoaneurysm, or urinary fistula, graded according to the Clavien-Dindo classification.
Console time | Perioperative/Periprocedural time
  Time in minutes from docking to undocking of the robotic system.
Length of hospital stay | From the date of surgery until the date of hospital discharge, assessed up to 30 days postoperatively
  Number of days from the date of surgery until the date of hospital discharge.
Participants requiring intraoperative conversion | Perioperative/Periprocedural time
  Number of participants converted to open or radical nephrectomy during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Nilo J Leão, MD., Principal Investigator — Brazilian Institute of Robotic Surgery
Locations (2):
- Brazil (2):
  - Hospital MaterDei Salvador, Salvador, Estado de Bahia
  - Brazilian Institute of Robotic Surgery, Salvador, Estado de Bahia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared in order to protect patient confidentiality and privacy. As the data may contain sensitive personal health information, maintaining strict confidentiality is essential and aligns with ethical and legal standards.

REFERENCES:
- [Background] Williams RD, Snowden C, Frank R, Thiel DD. Has Sliding-Clip Renorrhaphy Eliminated the Need for Collecting System Repair During Robot-Assisted Partial Nephrectomy? J Endourol. 2017 Mar;31(3):289-294. doi: 10.1089/end.2016.0562. Epub 2017 Jan 16. PMID 27960537
- [Background] Arora S, Bronkema C, Porter JR, Mottrie A, Dasgupta P, Challacombe B, Rha KH, Ahlawat RK, Capitanio U, Yuvaraja TB, Rawal S, Moon DA, Sivaraman A, Maes KK, Porpiglia F, Gautam G, Turkeri L, Bhandari M, Jeong W, Menon M, Rogers CG, Abdollah F. Omission of Cortical Renorrhaphy During Robotic Partial Nephrectomy: A Vattikuti Collective Quality Initiative Database Analysis. Urology. 2020 Dec;146:125-132. doi: 10.1016/j.urology.2020.09.003. Epub 2020 Sep 15. PMID 32941944
- [Background] Alrishan Alzouebi I, Williams A, Thiagarjan NR, Kumar M. Omitting Cortical Renorrhaphy in Robot-Assisted Partial Nephrectomy: Is it Safe? A Single Center Large Case Series. J Endourol. 2020 Aug;34(8):840-846. doi: 10.1089/end.2020.0121. PMID 32316759
- [Background] Bahler CD, Dube HT, Flynn KJ, Garg S, Monn MF, Gutwein LG, Mellon MJ, Foster RS, Cheng L, Sandrasegaran MK, Sundaram CP. Feasibility of omitting cortical renorrhaphy during robot-assisted partial nephrectomy: a matched analysis. J Endourol. 2015 May;29(5):548-55. doi: 10.1089/end.2014.0763. Epub 2015 Mar 10. PMID 25616087
- [Background] Kazama A, Attawettayanon W, Munoz-Lopez C, Rathi N, Lewis K, Maina E, Campbell RA, Lone Z, Boumitri M, Kaouk J, Haber GP, Haywood S, Almassi N, Weight C, Li J, Campbell SC. Parenchymal volume preservation during partial nephrectomy: improved methodology to assess impact and predictive factors. BJU Int. 2024 Aug;134(2):219-228. doi: 10.1111/bju.16300. Epub 2024 Feb 14. PMID 38355293
- [Background] Hung AJ, Cai J, Simmons MN, Gill IS. "Trifecta" in partial nephrectomy. J Urol. 2013 Jan;189(1):36-42. doi: 10.1016/j.juro.2012.09.042. Epub 2012 Nov 16. PMID 23164381
- [Background] Ruiz Guerrero E, Claro AVO, Ledo Cepero MJ, Soto Delgado M, Alvarez-Ossorio Fernandez JL. Robotic versus Laparoscopic Partial Nephrectomy in the New Era: Systematic Review. Cancers (Basel). 2023 Mar 16;15(6):1793. doi: 10.3390/cancers15061793. PMID 36980679
- [Background] Young M, Jackson-Spence F, Beltran L, Day E, Suarez C, Bex A, Powles T, Szabados B. Renal cell carcinoma. Lancet. 2024 Aug 3;404(10451):476-491. doi: 10.1016/S0140-6736(24)00917-6. Epub 2024 Jul 18. PMID 39033764
- [Background] Shatagopam K, Bahler CD, Sundaram CP. Renorrhaphy techniques and effect on renal function with robotic partial nephrectomy. World J Urol. 2020 May;38(5):1109-1112. doi: 10.1007/s00345-019-03033-w. Epub 2019 Dec 2. PMID 31792576
- [Background] Rose TL, Kim WY. Renal Cell Carcinoma: A Review. JAMA. 2024 Sep 24;332(12):1001-1010. doi: 10.1001/jama.2024.12848. PMID 39196544
- [Background] Makino T, Kadomoto S, Izumi K, Mizokami A. Epidemiology and Prevention of Renal Cell Carcinoma. Cancers (Basel). 2022 Aug 22;14(16):4059. doi: 10.3390/cancers14164059. PMID 36011051
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT07190638/Prot_SAP_000.pdf